CLINICAL TRIAL: NCT00977353
Title: N-methylglycine (Sarcosine) for Treatment of Major Depressive Disorder
Brief Title: N-methylglycine (Sarcosine) Treatment for Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Hsien-Yuan Lane, M.D., Ph.D, Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DOH95-TD-B-111-TM002
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Major Depressive Disorder; Depression; Major Depression
Keywords: Major depressive disorder; Depression; Sarcosine; N-methylglycine; NMDA
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Citalopram; Sarcosine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sarcosine (Experimental): sarcosine
  Interventions: Drug: sarcosine
- citalopram (Active Comparator): citalopram
  Interventions: Drug: citalopram

INTERVENTIONS:
Drug: citalopram — 20-60 mg/day, oral, for 6 weeks
  Arms: citalopram
Drug: sarcosine — 500-1500 mg/day, oral, for 6 weeks
  Arms: sarcosine

SUMMARY:
Major depressive disorder is a complex disease and most currently available antidepressants aiming at monoamine neurotransmission exhibit limited efficacy and cognitive effects. N-methyl-D-aspartate (NMDA), one subtype of glutamate receptors, plays an important role in learning and memory. N-methyl-D-aspartic acid (NMDA) enhancing agents, such as sarcosine (N-methylglycine), have been used as adjunctive therapy of schizophrenia. Sarcosine improved not only psychotic but also depressive symptoms in patients with schizophrenia. To confirm its antidepressant effect, the purpose of this study is to compare citalopram and sarcosine in efficacy for major depressive patients.

DETAILED DESCRIPTION:
Major depressive disorder is a complex disease and most currently available antidepressants aiming at monoamine neurotransmission exhibit limited efficacy and cognitive effects. Novel therapies via manipulating other neurotransmission (e.g. glutamate receptor) are being developed.

NMDA enhancing agents, such as sarcosine have been demonstrated to improve negative symptoms and depressive symptoms of schizophrenic patients. The purpose of this study is to compare citalopram and sarcosine in aspects of efficacy, safety in major depressive patients.

In the study, 40 major depressive patients are recruited into the 6-week trial and randomly assigned into the two groups (20-60 mg/d citalopram, or 500 - 1500 mg/d sarcosine) with a double-blind manner. Hamilton Depression Rating Scale(17-item), CGI(Clinical Global Impression), GAF(Global Assessment of Function)and side effects are evaluated every two weeks during the trial. The efficacies of two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years
* Fulfilled the DSM-IV criteria of major depressive disorder
* Had a 17-item Hamilton Rating Scale for Depression (HAMD-17)>or= 18
* No DSM-IV diagnosis of substance abuse or dependence (including alcohol) within the past 6 months
* Had been drug free for > 3 months
* Physically healthy and had all laboratory parameters within normal limits.
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* Had history of epilepsy, head trauma or other major neurological or medical diseases
* Had psychotic depression, bipolar I/II disorder, schizophrenia or any other psychotic disorder
* Moderate-severe suicidal risks
* Severe cognitive impairment
* Female subjects who were pregnant, or at risk of pregnancy or lactation
* Initiating or stopping formal psychotherapy within six weeks prior to enrollment
* Had a history of poor response to SSRIs or previously received electroconvulsive therapy
* Had a history of severe adverse reaction to SSRIs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Depression Rating Scale | week 0, 2, 4, 6
  score change
Remission rate | week 0, 2,4, 6
GAF(Global Assessment of Function) | Week 0, 2, 4, 6
  score changes

SECONDARY OUTCOMES:
dropout rate | week 0, 2, 4, 6
CGI(clinical global impression) | week 0, 2, 4,6
  score changes
Response Rate | Week 0, 2, 4, 6
Factors of 17-item Hamilton Depression Rating Scale | Week 0, 2, 4, 6

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Yuan Lane, M.D., Ph.D, Principal Investigator — Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan; Chieh-Liang Huang, MD, Principal Investigator — Department of Psychiatry, China Medical University Hospital,Taichung,Taiwan
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Huang CC, Wei IH, Huang CL, Chen KT, Tsai MH, Tsai P, Tun R, Huang KH, Chang YC, Lane HY, Tsai GE. Inhibition of glycine transporter-I as a novel mechanism for the treatment of depression. Biol Psychiatry. 2013 Nov 15;74(10):734-41. doi: 10.1016/j.biopsych.2013.02.020. Epub 2013 Apr 3. PMID 23562005